CLINICAL TRIAL: NCT02983045
Title: A Phase 1/2, Open-label, Multicenter Study of the Combination of NKTR-214 and Nivolumab or the Combination of NKTR-214, Nivolumab, and Other Anti-Cancer Therapies in Patients With Select Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: A Dose Escalation and Cohort Expansion Study of NKTR-214 in Combination With Nivolumab and Other Anti-Cancer Therapies in Patients With Select Advanced Solid Tumors
Acronym: PIVOT-02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-214-02
Record Dates: First submitted 2016-11-23; First posted 2016-12-06 (Estimated); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Melanoma; Renal Cell Carcinoma; Non Small Cell Lung Cancer; Urothelial Carcinoma; Triple Negative Breast Cancer; HR+/HER2- Breast Cancer; Gastric Cancer
Keywords: NKTR-214; Bempegaldesleukin; Nivolumab; Paclitaxel; Carboplatin; Cisplatin; Pemetrexed; Melanoma; Renal Cell Carcinoma; Non Small Cell Lung Cancer; Urothelial Carcinoma; Triple Negative Breast Cancer; HR+/HER2- Breast Cancer; Gastric Cancer; Colorectal Cancer; Metastatic; Advanced; Immunotherapy; Anti-PD-1; anti-CTLA-4
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Triple Negative Breast Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; bempegaldesleukin; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation: Combination of NKTR-214 + nivolumab (Experimental): NKTR 214 + nivolumab at 5 dosage levels to determine the RP2D Part 1 of RP2D in patients with advanced or metastatic melanoma, RCC, NSCLC, urothelial carcinoma, or TNBC.
  Interventions: Drug: Dose Escalation Doublet: Combination of NKTR-214 + nivolumab
- Dose Expansion: Combination of NKTR-214 + nivolumab (Experimental): NKTR-214+nivolumab in patients with advanced or metastatic solid tumor malignancies to assess the efficacy of the RP2D.
  Interventions: Drug: Dose Expansion Doublet: Combination of NKTR-214 + nivolumab
- Experimental: Combination of NKTR-214 + nivolumab + ipilimumab (Experimental): To assess the safety and tolerability of NKTR 214 + nivolumab + ipilimumab triplet therapy and establish RP2D dosing schedules for Part 4 in patients with advanced or metastatic melanoma, RCC, NSCLC, or UCC in a first-line setting (1L).
  Interventions: Drug: Schedule Finding Triplet: Combination of NKTR-214+ nivolumab+ ipilimumab
- Experimental: Dose Expansion of Part 3 (Experimental): To further assess the RP2D triplet combination dosing schedules from Part 3 in 1L NSCLC and 1L RCC patients.
  Interventions: Drug: Dose Expansion Triplet: Combination of NKTR-214+ nivolumab+ ipilimumab

INTERVENTIONS:
Drug: Dose Escalation Doublet: Combination of NKTR-214 + nivolumab — NKTR 214 + nivolumab at 5 dosage levels.
  Other Names: Bempegaldesleukin + Opdivo®
  Arms: Dose Escalation: Combination of NKTR-214 + nivolumab
Drug: Dose Expansion Doublet: Combination of NKTR-214 + nivolumab — Select patient cohorts with select tumor types will be dosed with NKTR-214 + nivolumab at the RP2D + other anti-cancer therapies per institution standard.
  Other Names: Bempegaldesleukin+ Opdivo®; Carboplatin (Paraplatin®); Cisplatin (Platinol®); Pemetrexed (Alimta®); Paclitaxel (Taxol®)
  Arms: Dose Expansion: Combination of NKTR-214 + nivolumab
Drug: Schedule Finding Triplet: Combination of NKTR-214+ nivolumab+ ipilimumab — 1L patients with RCC, NSCLC, UCC, and melanoma received NKTR-214 0.006 mg/kg q3w in combination with nivolumab and ipilimumab according to 3 dosing schedules.
  Other Names: Bempegaldesleukin+ Opdivo®+ Yervoy®
  Arms: Experimental: Combination of NKTR-214 + nivolumab + ipilimumab
Drug: Dose Expansion Triplet: Combination of NKTR-214+ nivolumab+ ipilimumab — Combination of NKTR-214 + nivolumab + ipilimumab was administered at RP2D dose/schedules in select tumor types
  Other Names: Bempegaldesleukin+ Opdivo®+ Yervoy®
  Arms: Experimental: Dose Expansion of Part 3

SUMMARY:
In this four-part study, NKTR-214 was administered in combination with nivolumab and with/without other anticancer therapies. Part 1 considered escalating doublet (NKTR 214 + nivolumab) doses to determine the RP2D. Part 2 considered dose expansion cohorts for the doublet (NKTR 214 + nivolumab ± chemotherapy). Part 3 was schedule-finding for a triplet therapy (NKTR 214 + nivolumab + ipilimumab). Part 4 dose expansion for the triplet (NKTR 214 + nivolumab + ipilimumab) was planned to further assess the efficacy of the RP2D triplet combination at dosing schedules from Part 3.

DETAILED DESCRIPTION:
Part 1 enrolled patients with advanced or metastatic melanoma, renal cell carcinoma (RCC), non-small cell lung cancer (NSCLC), urothelial carcinoma, or triple negative breast cancer (TNBC) to determine the recommended Phase 2 dose (RP2D) or maximum tolerated dose (MTD) of NKTR 214 + nivolumab doublet therapy.

Part 2 enrolled patients with advanced or metastatic solid tumor malignancies (including 9 tumor types consisting of the same 5 tumor types as in Part 1, plus hormone receptor positive human epidermal growth factor receptor 2 [HER 2] negative breast cancer [HR+ HER2- BC], gastric cancer, colorectal carcinoma, and small cell lung cancer [SCLC]) to assess the efficacy of the RP2D.

Part 3 enrolled patients with advanced or metastatic melanoma, RCC, NSCLC, or urothelial carcinoma (UCC) in a first-line setting (1L) to assess the safety and tolerability of NKTR 214 + nivolumab + ipilimumab triplet therapy Three dosing schedules were evaluated to establish RP2D dosing schedules for Part 4 of the study.

Part 4 planned to enroll patients with advanced or metastatic melanoma, RCC, NSCLC, or UCC to further assess the efficacy of the RP2D triplet combination at the 3 dosing schedules from Part 3. Patients were enrolled simultaneously to each tumor cohort.

All patients enrolled in the study were closely monitored for safety, tolerability and response per RECIST criteria. The primary efficacy endpoint was objective response rate (ORR) using RECIST 1.1 at the RP2D doublet.

ELIGIBILITY:
INCLUSION CRITERIA - For Parts 1-4:

* Histologically confirmed diagnosis of a locally advanced (not amenable to curative therapy such as surgical resection) or metastatic solid tumors
* Life expectancy > 12 weeks
* Patients must not have received prior interleukin-2 (IL-2) therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Measurable disease per RECIST 1.1
* Patients with stable brain metastases under certain criteria
* Fresh and archival tumor tissue available Tumor specific inclusion criteria may apply.

EXCLUSION CRITERIA - For Parts 1-4:

* Use of an investigational agent or an investigational device within 28 days before administration of first dose of NKTR--214
* Females who are pregnant or breastfeeding
* Participants who have an active autoimmune disease requiring systemic treatment within the past 3 months or have a documented history of clinically severe autoimmune disease that requires systemic steroids or immunosuppressive agents
* History of organ transplant that requires use of immune suppressive agents
* Active malignancy not related to the current diagnosed malignancy
* Evidence of clinically significant interstitial lung disease or active, noninfectious pneumonitis
* Participants who have had < 28 days since the last chemotherapy, biological therapy, or < 14 days from approved tyrosine kinase inhibitor (TKI) therapy, or systemic or inhaled steroid therapy at doses greater than 10mg of prednisone Tumor specific exclusion criteria may apply.

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (58):
- United States (22):
  - UCSD, Moores Cancer Center, La Jolla, California
  - UCLA, Los Angeles, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado, Denver, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Orlando Health Inc., Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Chicago, Maywood, Illinois
  - Indiana University Health Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center - NYU Cancer Institute, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (5):
  - Antwerp University Hospital, Edegem
  - Vzw Az Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - GZA Ziekenhuizen Campus Sint-Augustinus, Wilrijk
- Canada (4):
  - BC Cancer Agency Vancouver Centre, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (5):
  - L'Institut Paoli - Calmettes, Marseille, Brouches-duRhone
  - Institut de Cancerologie de l'Ouest, Saint-Herblain, Loire-Atlantique
  - Centre Léon Bérard, Lyon
  - Assistance Publique Hopitaux de Marseille - Hopital Nord, Marseille
  - Gustave Roussy, Villejuif
- Italy (6):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Institute for Cancer Research and Treatment (IRCC), Turin
- Poland (6):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny im. Ks. B. Markiewicza, Brzozów
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Instytut Medyczny Santa Familia Sp. z o. o. w Łodzi, Lodz
  - Mazowieckie Centrum Leczenia Chorób Płuc i Gruźlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii, Poznan
  - Med-Polonia Sp. z o.o., Poznan
- Spain (7):
  - Hospital Quirón Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Campus Hospital Universitario Virgen del Rocío - Instituto de Biomedicina de Sevilla (IBIS), Seville
- United Kingdom (3):
  - The Royal Marsden NHS Trust, London
  - Mount Vernon Cancer Centre, Northwood
  - The Christie NHS Foundation Trust, Withington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siefker-Radtke AO, Cho DC, Diab A, Sznol M, Bilen MA, Balar AV, Grignani G, Puente E, Tang L, Chien D, Hoch U, Choudhury A, Yu D, Currie SL, Tagliaferri MA, Zalevsky J, Hurwitz ME, Tannir NM. Bempegaldesleukin plus Nivolumab in First-line Metastatic Urothelial Carcinoma: Results from PIVOT-02. Eur Urol. 2022 Oct;82(4):365-373. doi: 10.1016/j.eururo.2022.05.002. Epub 2022 May 25. PMID 35643589
- [Derived] Diab A, Tykodi SS, Daniels GA, Maio M, Curti BD, Lewis KD, Jang S, Kalinka E, Puzanov I, Spira AI, Cho DC, Guan S, Puente E, Nguyen T, Hoch U, Currie SL, Lin W, Tagliaferri MA, Zalevsky J, Sznol M, Hurwitz ME. Bempegaldesleukin Plus Nivolumab in First-Line Metastatic Melanoma. J Clin Oncol. 2021 Sep 10;39(26):2914-2925. doi: 10.1200/JCO.21.00675. Epub 2021 Jul 13. PMID 34255535
- [Derived] Veatch JR, Singhi N, Jesernig B, Paulson KG, Zalevsky J, Iaccucci E, Tykodi SS, Riddell SR. Mobilization of pre-existing polyclonal T cells specific to neoantigens but not self-antigens during treatment of a patient with melanoma with bempegaldesleukin and nivolumab. J Immunother Cancer. 2020 Dec;8(2):e001591. doi: 10.1136/jitc-2020-001591. PMID 33298619

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 240 mg nivolumab q2w.
- Part 1 Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.006 mg/kg administered every 2 weeks (q2w) in combination with 240 mg nivolumab q2w.
- Part 1 Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.003 mg/kg administered every 2 weeks (q2w) in combination with 240 mg nivolumab q2w.
- Part 1 Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
- Part 1 Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.009 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
- Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w: In this Part 2 of the study, the patients will receive a combination of NKTR-214 + nivolumab at the RP2D (NKTR 214 0.006 mg/kg q3w + nivolumab 360 mg q3w) with or without chemotherapy.
- Part 3 Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab: In this Part 3 of the study, patients will receive a combination of NKTR-214 at 0.006 mg/kg q3w with nivolumab and ipilimumab in up to three different dosing schedules to identify dose and schedules that proceed into Part 4.
  In Schedule 1, patients received NKTR-214 at 0.006 mg/kg q3w + nivolumab at 360 mg flat dose q3w + ipilimumab at 1 mg/kg q6w.
- Part 3 Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab: In this Part 3 of the study, patients will receive a combination of NKTR-214 at 0.006 mg/kg q3w with nivolumab and ipilimumab in up to three different dosing schedules to identify dose and schedules that proceed into Part 4.
  In Schedule 2, patients received NKTR-214 at 0.006 mg/kg q3w + nivolumab at 1 mg/kg q3w + ipilimumab at 3 mg/kg q3w for four cycles, followed by the maintenance dose of NKTR-214 0.006 mg/kg and nivolumab 360 mg q3w.
- Part 3 Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab: In this Part 3 of the study, patients will receive a combination of NKTR-214 at 0.006 mg/kg q3w with nivolumab and ipilimumab in up to three different dosing schedules to identify dose and schedules that proceed into Part 4.
  In Schedule 3, patients received NKTR-214 at 0.006 mg/kg q3w + nivolumab at 3 mg/kg q3w + ipilimumab at 1 mg/kg q3w for four cycles, followed by the maintenance dose of NKTR-214 0.006 mg/kg and nivolumab 360 mg q3w.
- Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab: Experimental Combination of NKTR-214 + nivolumab + ipilimumab
  Combination of NKTR-214 + nivolumab: Combination of NKTR-214 + nivolumab +ipilimumab administered at the RP2D dose/schedule.
Period: Overall Study
Arm/Group | Part 1 Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 1 Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 3 Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab | Part 3 Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab | Part 3 Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab | Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab
Started | 4 | 3 | 3 | 25 | 3 | 476 | 10 | 8 | 6 | 19
Completed | 4 | 2 | 3 | 20 | 3 | 394 | 10 | 8 | 6 | 17
Not Completed | 0 | 1 | 0 | 5 | 0 | 82 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 5 | 0 | 72 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab: Experimental Combination of NKTR-214 + nivolumab ipilimumab that may enroll between 12-26 patients per tumor type
  Combination of NKTR-214 + nivolumab: Combination of NKTR-214 + nivolumab +ipilimumab administered at the RP2D dose/schedule.
- Total: Total of all reporting groups
Arm/Group | Part 1 Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 1 Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 3 Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab | Part 3 Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab | Part 3 Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab | Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 4 | 3 | 3 | 25 | 3 | 476 | 10 | 8 | 6 | 19 | 557
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.90) | 61.7 (7.37) | 57.0 (7.81) | 59.2 (10.12) | 55.7 (6.81) | 62.1 (11.48) | 62.4 (9.45) | 64.3 (5.85) | 61.2 (9.3) | 59.1 (12.63) | 61.7 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 5 | 1 | 207 | 1 | 0 | 0 | 5 | 221
  Male | 2 | 3 | 3 | 20 | 2 | 269 | 9 | 8 | 6 | 14 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 2 | 35 | 1 | 2 | 2 | 2 | 46
  Not Hispanic or Latino | 4 | 3 | 1 | 24 | 1 | 413 | 9 | 6 | 4 | 15 | 480
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 28 | 0 | 0 | 0 | 2 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 16 | 1 | 1 | 0 | 0 | 20
  White | 4 | 3 | 3 | 23 | 3 | 413 | 8 | 7 | 5 | 17 | 486
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 31 | 1 | 0 | 1 | 2 | 35
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 0 | 0 | 27 | 0 | 0 | 0 | 0 | 27
  Belgium | 0 | 0 | 0 | 0 | 0 | 29 | 0 | 0 | 0 | 0 | 29
  United States | 4 | 3 | 3 | 25 | 3 | 295 | 10 | 8 | 6 | 19 | 376
  Poland | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 23
  Italy | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0 | 35
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 6
  France | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 14
  Spain | 0 | 0 | 0 | 0 | 0 | 47 | 0 | 0 | 0 | 0 | 47
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status:
  ECOG Performance Status of 0 = Able to carry out all normal activities without restriction
  ECOG Performance Status of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature
  Participants
    0 | 3 | 2 | 2 | 16 | 3 | 221 | 6 | 6 | 5 | 12 | 276
    1 | 1 | 1 | 1 | 9 | 0 | 254 | 4 | 2 | 1 | 7 | 280
    Data Missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1 Dose Escalation: Incidence of Dose-limiting Toxicity (DLT) During the DLT Evaluation Window
Description: Part 1of the study was a dose-escalation phase that evaluated the safety and tolerability and defined the maximum tolerated dose or recommended Phase 2 dose of the NKTR-214/nivolumab doublet across 5 dosage/schedule levels. The results presented are for the DLT Population.
Time Frame: Includes DLTs that occurred within the DLT window of at least 21 days after the first dose of study treatment (28 days for every 2 weeks dosing; 21 days for every 3 weeks dosing). Patients were counted only once under each preferred term.
Population: The DLT population included all Part 1 patients who took study treatment and followed up at least through the DLT evaluation period (q2w dosing: received ≥ 2 cycles of study treatment and stayed in study for at least 28 days; q3w dosing: received at least 1 cycle of study treatment and stayed in study for at least 21 days) or discontinued from study treatment due to DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 240 mg nivolumab q2w.
- Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.006 mg/kg administered every 2 weeks (q2w) in combination with 240 mg nivolumab q2w.
- Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.003 mg/kg administered every 2 weeks (q2w) in combination with 240 mg nivolumab q2w.
- Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.006 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
- Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w: NKTR-214 in escalating doses combined with one of the two proposed doses of nivolumab. The goal of this dose escalation Part 1 of the study is to find the RP2D.
  Patients will receive NKTR-214 at 0.009 mg/kg administered every 3 weeks (q3w) in combination with 360 mg nivolumab q3w.
Arm/Group | Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w | Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w | Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w | Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w
Number analyzed (Participants) | 4 | 3 | 3 | 24 | 3
Participants
  At least 1 DLT | 0 | 0 | 0 | 0 | 2
  Metabolism and Nutrition Disorders: Acidosis | 0 | 0 | 0 | 0 | 1
  Metabolism and Nutrition Disorders: Hyperglycaemia | 0 | 0 | 0 | 0 | 1
  Vascular Disorders: Hypotension | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Part 3 Schedule Finding: Incidence of Dose-limiting Toxicity (DLT) During the DLT Evaluation Window
Description: Part 3 of the study was a schedule finding phase to establish the recommended phase 2 dosing schedules for Part 4 and assess the safety and tolerability for the NKTR-214/nivolumab/ipilimumab triplet combination. The results presented are for the DLT Population.
Time Frame: Dose-limiting toxicities (DLTs) were assessed during a 3-week (21-day) DLT evaluation period beginning with the first dose of ipilimumab.
Population: The DLT population included all Part 3 patients who received at least 1 cycle of study treatment and stayed in study for at least 21 days after first dose of ipilimumab or discontinued from study treatment due to DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab: In this Part 3 of the study, patients will receive a combination of NKTR-214 at 0.006 mg/kg q3w with nivolumab and ipilimumab in up to three different dosing schedules to identify dose and schedules that proceed into Part 4.
  In Schedule 1, patients received NKTR-214 at 0.006 mg/kg q3w + nivolumab at 360 mg flat dose q3w + ipilimumab at 1 mg/kg q6w.
- Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab: In this Part 3 of the study, patients will receive a combination of NKTR-214 at 0.006 mg/kg q3w with nivolumab and ipilimumab in up to three different dosing schedules to identify dose and schedules that proceed into Part 4.
  In Schedule 2, patients received NKTR-214 at 0.006 mg/kg q3w + nivolumab at 1 mg/kg q3w + ipilimumab at 3 mg/kg q3w for four cycles, followed by the maintenance dose of NKTR-214 0.006 mg/kg and nivolumab 360 mg q3w.
- Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab: In this Part 3 of the study, patients will receive a combination of NKTR-214 at 0.006 mg/kg q3w with nivolumab and ipilimumab in up to three different dosing schedules to identify dose and schedules that proceed into Part 4.
  In Schedule 3, patients received NKTR-214 at 0.006 mg/kg q3w + nivolumab at 3 mg/kg q3w + ipilimumab at 1 mg/kg q3w for four cycles, followed by the maintenance dose of NKTR-214 0.006 mg/kg and nivolumab 360 mg q3w.
Arm/Group | Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab | Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab | Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 10 | 8 | 6
Participants
  Patients with at least one event | 1 | 1 | 1
  Endocrine disorders: Adrenal insufficiency | 0 | 1 | 0
  Endocrine disorders: Hyperthyroidism | 0 | 0 | 1
  Metabolism and nutrition disorders: Hyponatraemia | 1 | 0 | 0

3. Primary Outcome: Part 2 and Part 4: Objective Response Rate (ORR) Per RECIST 1.1 at Recommended Phase 2 Dose (RP2D)
Description: Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) at Recommended Phase 2 Dose (RP2D).
  ORR is defined as the percentage of enrolled participants who achieved a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR is calculated as the sum of CR and PR.
Time Frame: Tumor assessment at Screening then every 8 weeks (± 7 days) from Cycle 1 Day 1 and end of treatment (unless scan done within 4 weeks) up to approximately 27 months.
Population: The response evaluable population included patients who had measurable disease (per RECIST 1.1) at baseline and also had at least 1 postbaseline assessment of tumor response prior to receiving new systemic anticancer therapy, surgical procedures or radiotherapy on target lesions.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w: In this Part 2 of the study, the patients received a combination of NKTR-214 + nivolumab at the RP2D (NKTR 214 0.006 mg/kg q3w + nivolumab 360 mg q3w) with or without chemotherapy.
Arm/Group | Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 429 | 17
Participants | 64 | 3

ADVERSE EVENTS:
Time Frame: AEs were reported from the time of first study drug(s) administration until 100 days after the last dose of all study drug(s), up to a maximum of approximately 2.5 years.
Groups:
- Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab: Experimental Combination of NKTR-214 + nivolumab + ipilimumab. Combination of NKTR-214 + nivolumab: Combination of NKTR-214 + nivolumab +ipilimumab administered at the RP2D dose/schedule.
Arm/Group | Part 1 Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w | Part 1 Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 1 Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w | Part 3 Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab | Part 3 Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab | Part 3 Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab | Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/3 | 2/3 | 10/25 | 1/3 | 291/476 | 2/10 | 3/8 | 1/6 | 5/19
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 1/3 | 9/25 | 2/3 | 213/476 | 6/10 | 5/8 | 2/6 | 8/19
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 25/25 | 3/3 | 468/476 | 10/10 | 8/8 | 6/6 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w (N=4) | Part 1 Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w (N=3) | Part 1 Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w (N=3) | Part 1 Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w (N=25) | Part 1 Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w (N=3) | Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w (N=476) | Part 3 Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab (N=10) | Part 3 Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab (N=8) | Part 3 Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab (N=6) | Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab (N=19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bursitis infective staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 16 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 11 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 5 | 1 | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 15 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 7 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 0 | 1
Autoimmune nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Autoimmune hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Dose Escalation Cohort 1: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (240 mg) q2w (N=4) | Part 1 Dose Escalation Cohort 2: NKTR-214 (0.006 mg/kg) q2w + Nivolumab (240 mg) q2w (N=3) | Part 1 Dose Escalation Cohort 3: NKTR-214 (0.003 mg/kg) q2w + Nivolumab (240 mg) q2w (N=3) | Part 1 Dose Escalation Cohort 4: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w (N=25) | Part 1 Dose Escalation Cohort 5: NKTR-214 (0.009 mg/kg) q3w + Nivolumab (360 mg) q3w (N=3) | Part 2 Dose Expansion: NKTR-214 (0.006 mg/kg) q3w + Nivolumab (360 mg) q3w (N=476) | Part 3 Schedule Finding (Schedule 1): NKTR-214 + Nivolumab + Ipilimumab (N=10) | Part 3 Schedule Finding (Schedule 2): NKTR-214 + Nivolumab + Ipilimumab (N=8) | Part 3 Schedule Finding (Schedule 3): NKTR-214 + Nivolumab + Ipilimumab (N=6) | Part 4 Dose Expansion of NKTR-214 + Nivolumab + Ipilimumab (N=19)
Fatigue (General disorders) | 4 | 2 | 1 | 19 | 2 | 241 | 9 | 5 | 6 | 15
Pyrexia (General disorders) | 4 | 3 | 2 | 13 | 3 | 228 | 7 | 3 | 5 | 10
Influenza like illness (General disorders) | 3 | 0 | 0 | 14 | 1 | 126 | 6 | 6 | 6 | 13
Chills (General disorders) | 3 | 3 | 3 | 16 | 2 | 115 | 5 | 3 | 1 | 7
Oedema peripheral (General disorders) | 1 | 2 | 1 | 11 | 2 | 90 | 3 | 3 | 4 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 70 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 2 | 0 | 1 | 5 | 1 | 27 | 2 | 2 | 1 | 2
Malaise (General disorders) | 2 | 0 | 1 | 3 | 0 | 24 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 4 | 0 | 23 | 1 | 1 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 20 | 1 | 1 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 2 | 0 | 17 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 1 | 16 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 3 | 0 | 12 | 0 | 2 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 8 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 13 | 1 | 191 | 8 | 4 | 6 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 2 | 13 | 2 | 126 | 8 | 6 | 2 | 10
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 7 | 2 | 117 | 5 | 3 | 5 | 5
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 8 | 1 | 98 | 4 | 3 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 1 | 57 | 3 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 8 | 1 | 50 | 1 | 2 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 1 | 35 | 1 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 29 | 1 | 2 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 21 | 0 | 2 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 16 | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 14 | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 13 | 0 | 0 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 10 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 7 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 5 | 0 | 0 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 14 | 2 | 181 | 4 | 6 | 6 | 9
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 14 | 3 | 123 | 5 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 5 | 0 | 73 | 5 | 4 | 4 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 8 | 2 | 63 | 1 | 2 | 5 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 6 | 0 | 45 | 2 | 0 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3 | 0 | 23 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 18 | 1 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 17 | 0 | 2 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 16 | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 1 | 9 | 0 | 1 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 14 | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 13 | 0 | 1 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 8 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 8 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 15 | 2 | 118 | 4 | 4 | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 5 | 0 | 94 | 5 | 4 | 1 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 10 | 2 | 49 | 2 | 4 | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 5 | 2 | 34 | 0 | 0 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 5 | 0 | 24 | 0 | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 20 | 2 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 0 | 19 | 0 | 1 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 19 | 1 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 16 | 1 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 18 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 18 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 10 | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 10 | 1 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 1 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 14 | 1 | 114 | 2 | 2 | 5 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 9 | 0 | 80 | 2 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 9 | 0 | 68 | 2 | 0 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 5 | 0 | 45 | 0 | 1 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 2 | 30 | 3 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 28 | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0 | 19 | 1 | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 0 | 17 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 14 | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 11 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 9 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 9 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 0 | 12 | 2 | 168 | 4 | 4 | 6 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 41 | 2 | 2 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 23 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 19 | 1 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 17 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 8 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 7 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 1 | 1 | 12 | 1 | 73 | 2 | 2 | 3 | 6
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 7 | 1 | 79 | 2 | 3 | 3 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 5 | 1 | 32 | 1 | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 28 | 0 | 3 | 2 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 18 | 0 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 0 | 6 | 1 | 7 | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 13 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 5 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balint's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 3 | 1 | 64 | 2 | 1 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 30 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 18 | 2 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 16 | 1 | 0 | 2 | 1
Lipase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 13 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 13 | 1 | 0 | 1 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 9 | 0 | 77 | 3 | 2 | 2 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 31 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 3 | 2 | 1 | 2 | 0 | 20 | 0 | 2 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 10 | 0 | 1 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 35 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 3 | 0 | 28 | 3 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 2 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 6 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis pseudomonas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 5 | 1 | 51 | 3 | 1 | 3 | 5
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 16 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 7 | 1 | 65 | 2 | 5 | 2 | 5
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 25 | 0 | 3 | 1 | 2
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 0 | 1
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 12 | 2 | 1 | 0 | 4
Vision blurred (Eye disorders) | 1 | 1 | 0 | 4 | 0 | 12 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 9 | 1 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 2 | 0 | 5 | 1 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3 | 0 | 29 | 1 | 1 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 51 | 0 | 0 | 0 | 4
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 9 | 1 | 0 | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 11 | 1 | 1 | 1 | 5
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 17 | 1 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 10 | 2 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 9 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 13 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 11 | 1 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 7 | 1 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 7 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 9 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 8 | 0 | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT02983045/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT02983045/SAP_001.pdf